CLINICAL TRIAL: NCT05506527
Title: Assessment of Respiratory Function in Children With Cerebral Palsy Using Combined Plyometric Exercise and Sensorimotor Program: A Randomized Controlled Trial
Brief Title: Assessment of Respiratory Function Cerebral Palsy Using Plyometric Exercise Sensorimotor Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Egyptian Chinese University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelmoneim El Meligy, lecturer of physical therapy for pediatrics, Egyptian Chinese University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003787
Record Dates: First submitted 2022-08-15; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Cerebral Palsy
Keywords: respiratory capacity; cerebral palsy; plyometric exercise
MeSH Terms: conditions — Cerebral Palsy | interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Participant
Masking Description: lottery method
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group 1 (Experimental): Study group A: will receive combined plyometric exercises and sensorimotor program
  Interventions: Other: Sensorimotor program and plyometric exercise
- study group 2 (Experimental): Study group B: will receive sensorimotor program alone
  Interventions: Other: Sensorimotor program and plyometric exercise

INTERVENTIONS:
Other: Sensorimotor program and plyometric exercise — Children in study group A will receive combined plyometric exercises (vertical paradigm) and sensorimotor program
  - Children of the study group B will receive sensorimotor program alone.

SUMMARY:
To examine if adding plyometric exercises to sensorimotor exercises would improve respiratory function in children and adolescents with cerebral palsy

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a varied group of developmental disorders secondary to a static immature brain injury that primarily results in persistent nonspecific impairment of movement and posture. Approximately 25% of all CP cases experience disturbance of motor function with unilateral spasticity pertaining to the upper and lower extremities contralateral to the affected cerebral hemisphere and categorized as spastic hemiplegia. Some asymmetries might be noted when hemiplegic children are attempting to perform motor activities. In supported standing, hemiplegic children may stand preferentially on their more functional side and exhibit postural malalignments that impair the ability to transfer body weight on the affected lower extremity.

Children and adolescents with CP have poor respiratory function, secondary to the disease process. Impaired airway clearance, recurrent aspirations, chest infections, poor cough mechanism, impaired lung function, deformity of the spine and chest, and poor nutrition status influence the respiratory condition of children and adults with CP resulting in reduced lung capacity in these individuals.

Plyometric exercises are a specific pattern of resistive strength training in which the muscle starts to contract eccentrically followed by rapid concentric contraction of the same muscle. It can jointly generate high velocity dynamic movements and high-impact force on the muscles and bones. Currently, a limited number of studies have analysed the efficacy of the plyometric training on respiratory function in children with CP or any other disabling health conditions. Preliminary studies have demonstrated the positive effect of plyometric exercises for the gross motor function in boys with unilateral CP.

ELIGIBILITY:
Inclusion Criteria:

* Age will be 8 - 14 years.
* children will be assigned to the study are suffering from spastic hemiplegic cerebral palsy (less than grade 1+ om Modified Ashwar Scale)
* Considering the physical problems, children will be chosen according to Growth Motor Function Classification System (GMFCS) with levels I-III
* The ability to understand simple verbal instructions.

Exclusion Criteria:

* Visual and hearing impairment; surgery within the last three months preventing them from taking part in sensorimotor physical therapy
* Severe oromotor issues
* Severe chest infections

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
change of spasticity | six weeks
  will be measured by modified Ashower Scale

SECONDARY OUTCOMES:
change of Respiratory capacity and vital capacity | six weeks
  will be measured by incentive spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Eman Abdel-Halim, Study Director — Cairo University
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No